CLINICAL TRIAL: NCT03933436
Title: EPIC: Effect of Povidone Iodine Periurethral Cleansing on Level of Contamination With Clean Catch: A Randomized Control Trial
Brief Title: EPIC: Effect of Povidone Iodine Periurethral Cleansing on Level of Contamination With Clean Catch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Travis Callahan (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Travis Callahan, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FWH20190009H
Record Dates: First submitted 2019-04-23; First posted 2019-05-01 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Urine Contamination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iodine (Experimental): Iodine swabs.
  Interventions: Other: Iodine swabs.
- Normal Saline (Active Comparator): Saline flush.
  Interventions: Other: Saline flush.

INTERVENTIONS:
Other: Iodine swabs. — Children will then have their periurethral region gently cleansed for ten seconds with iodine swabs.
  Arms: Iodine
Other: Saline flush. — Children will then have their periurethral region gently cleansed for ten seconds with saline flush.
  Arms: Normal Saline

SUMMARY:
The primary aim of this study is to see if the use of an antiseptic preparation (povidone iodine) versus cold normal saline, will decrease rates of urine contamination during the non-invasive Quick Wee (QW) collection of pediatric urine.

DETAILED DESCRIPTION:
Urinary tract infections (UTI) are common acute illnesses among pediatric patients, accounting for 5-7% of emergency department visits in the under two-year-old population. However, obtaining urine samples from the precontinent patient can be difficult. There is an ongoing debate regarding which noninvasive method for urine specimen collection is best for this population. The main argument against clean catch is the high rate of contamination compared to invasive collection and reliability.

There are many methods of noninvasive urine collection. These methods are preferred as they are fairly well tolerated by patients, less distressing to parents, cost effective, and require less technical expertise. In the past; these methods have been dismissed due to their high rates of contamination, time to void and also effectiveness. The National Institute of Health and Clinical Excellence (NICE, UK) recommends a clean-catch urine (CCU) be the first attempt at obtaining a urine specimen from children suspected of having UTI. This means placing the urine specimen collection container into the urine mid-stream once the child has begun to void to avoid contamination. Conversely, the American Academy of Pediatrics recommends clean catch urine for screening and a catheter specimen urine collection or suprapubic aspiration for definitive diagnosis. Both of these invasive techniques produce quick urine samples with low rates of contamination; however they can be painful and distressing to both the patient and parent.

The Quick-Wee method for noninvasive urine collection has been evaluated in a one randomized controlled trial and has been shown to significantly increase the five minute voiding success rate for CC urine collection; 31%, n= 174. However a past study demonstrated contamination rate of 27%, n=174. No study has directly evaluated the use of antiseptic solution in the evaluation of the QW rate of contamination in pediatric patients. The purpose of this study is to see whether the use of povidone iodine swabs prior to the QW method will decrease the rate of contamination. A decrease of the rate of contamination would strengthen the validity of this simple CCU method. Also using the this method for the collection method in both the experimental and control groups will further evaluated the five min void success rate.

The investigators chose to use iodine as the prepping agent because it is currently the standard cleaning solution used for adult and pediatric patients. It is readily available, inexpensive and has been shown to be less caustic then other prepping agents.

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* DoD children aged one month (28 days) to 12 months (365 days) (if the child was born less than 36 weeks gestation, age will be corrected)
* Precontinent (meaning that the child is unable to void on command)
* Treating clinician has determined that the child requires urine sample collection for course of treatment.

Exclusion Criteria:

* If the treating clinician has determined that there is a need for immediate treatment and urine sample collection via invasive method, any type of anatomical or neurologic condition that will affect the ability to void or sensation of the suprapubic area.
* Children with past hypersensitivity reactions to iodine swabs.

Ages: 28 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Number of participant samples indicating urine contamination | 24 to 48 hours
  Binary yes/no outcome of detection of microbial markers to determine level of contamination

SECONDARY OUTCOMES:
Number of participants who void urine | 5 minutes
  Binary yes/no outcome of voiding urine

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Crawford, MD, Study Director — Mike O'Callaghan Military Medical Center, 99MDG, US Air Force
Locations (1):
- Mike O'Callaghan Military Medical Center, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaw KN, Gorelick M, McGowan KL, Yakscoe NM, Schwartz JS. Prevalence of urinary tract infection in febrile young children in the emergency department. Pediatrics. 1998 Aug;102(2):e16. doi: 10.1542/peds.102.2.e16. PMID 9685461
- [Background] National Collaborating Centre for Women's and Children's Health (UK). Urinary Tract Infection in Children: Diagnosis, Treatment and Long-term Management. London: RCOG Press; 2007 Aug. Available from http://www.ncbi.nlm.nih.gov/books/NBK50606/ PMID 21290637
- [Background] Practice parameter: the diagnosis, treatment, and evaluation of the initial urinary tract infection in febrile infants and young children. American Academy of Pediatrics. Committee on Quality Improvement. Subcommittee on Urinary Tract Infection. Pediatrics. 1999 Apr;103(4 Pt 1):843-52. doi: 10.1542/peds.103.4.843. PMID 10103321

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT03933436/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT03933436/ICF_001.pdf